CLINICAL TRIAL: NCT01498952
Title: A Phase 1b/2, Open-label, Randomized Study of MEDI-573 in Combination With Sorafenib Verses Sorafenib Alone in Adult Subjects With Unresectable or Metastatic Hepatocellular Carcinoma
Brief Title: MEDI-573 in Combination With SOC in Unresectable or Metastatic HCC.
Acronym: MEDI-573-1028
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI-573-1028
Record Dates: First submitted 2011-11-29; First posted 2011-12-26 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Unresectable or Metastatic Hepatocellular Carcinoma (HCC)
Keywords: HCC, liver cancer, hepatocellular carcinoma, MEDI-573, anti-IGF
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — dusigitumab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1b Cohort A (Experimental): Participants will receive MEDI-573 10 mg/kg intravenous infusion on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573 (1 of 3 doses); Drug: Sorafenib
- Phase 1b Cohort B (Experimental): Participants will receive MEDI-573 45 mg/kg intravenous infusion on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573 (1 of 3 doses); Drug: Sorafenib
- Phase 1b Cohort C (Experimental): Participants will receive MEDI-573 30 mg/kg intravenous infusion on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573 (1 of 3 doses); Drug: Sorafenib
- Phase 2 Arm 1 (Experimental): Participants will receive recommended dose of MEDI-573 from Phase 1b IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
  Interventions: Drug: MEDI-573 (1 of 3 doses); Drug: Sorafenib
- Phase 2 Arm 2 (Active Comparator): Participants will receive sorafenib 400 mg orally twice daily until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: MEDI-573 (1 of 3 doses) — MEDI-573, a human immunoglobulin G2 lambda (IgG2λ) monoclonal antibody (MAb), is a dual-targeting human antibody that neutralizes insulin-like growth factor (IGF)-I and IGF-II ligands
  Arms: Phase 1b Cohort A; Phase 1b Cohort B; Phase 1b Cohort C; Phase 2 Arm 1
Drug: Sorafenib — Sorafenib is a tyrosine kinase inhibitor, anti-angiogenic, VEGF inhibitor

SUMMARY:
A Phase 1b/2, open-label, randomized study to evaluate MEDI-573 in combination with standard of care in adult subjects with unresectable or metastatic hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or minimum age of consent per local regulations at the time of screening
* Unresectable or metastatic hepatocellular carcinoma
* ECOG Performance Status ≤ 2
* Life expectancy of ≥ 3 months;

Exclusion Criteria:

* Child-Pugh Score for Cirrhosis Mortality > 7 points
* Prior or current system anti-cancer therapy for HCC, including cytotoxic, biologic, targeted or experimental therapy
* Prior local treatment for HCC less than 4 weeks prior to initiating study treatment
* Active second malignancy
* Major surgery, open biopsy or significant traumatic injury within 4 weeks prior to initiating study treatment
* Thrombotic or embolic events within 6 months prior to initiating study treatment
* Ongoing pancreatitis
* Uncontrolled or refractory ascites
* Evidence of ongoing spinal cord compression, known carcinomatous meningitis, or known leptomeningeal carcinomatosis
* Hepatic encephalopathy > Grade 1
* Active brain metastases with exceptions
* Poorly controlled diabetes mellitus
* Active coronary artery disease
* Uncontrolled hypertension

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2013-04-09 (Actual); Study Completion 2013-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perez, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Research Site, Oxnard, California
  - Research Site, Golden Springs, Colorado
  - Research Site, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the USA.
Pre-assignment Details: Phase 2 part of the study was not launched by the sponsor due to strategic business reasons. No participants were randomized in Phase 1b Cohort C part of the study as no dose limiting toxicity was observed in Phase 1b Cohort B.
Groups:
- Phase 1b Cohort A: Participants received MEDI-573 10 mg/kg intravenous infusion (IV) on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
- Phase 1b Cohort B: Participants received MEDI-573 45 mg/kg IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
- Phase 1b Cohort C: Participants were planned to receive MEDI-573 30 mg/kg IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
- Phase 2 Arm 1: Participants were planned to receive recommended dose of MEDI-573 from Phase 1b IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
- Phase 2 Arm 2: Participants were planned to receive sorafenib 400 mg orally twice daily until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
Period: Overall Study
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Phase 1b Cohort C | Phase 2 Arm 1 | Phase 2 Arm 2
Started | 3 | 3 | 0 | 0 | 0
Completed | 1 | 1 | 0 | 0 | 0
Not Completed | 2 | 2 | 0 | 0 | 0
Not completed — Death | 2 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any amount of study treatment.
Groups:
- Phase 1b Cohort A: Participants received MEDI-573 10 mg/kg IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily as background therapy until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.7 (1.2) | 65.7 (11.6) | 66.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The DLT was defined as any Grade 3 or higher hematologic or non-hematologic toxicity considered to be related to MEDI-573 that occurred during the DLT evaluation period (Days 1 to 21 of Cycle 1), with the exceptions of Grade 3 fever (occurred in the absence of neutropenia and resolved to normal or baseline within 24 hours of treatment and was not considered as SAE), Grade 3 rigors/chills that responded to optimal therapy, and Grade < 4 hyperglycemia that resolved in < 24 hours.
Time Frame: Day 1 to Day 21 of Cycle 1
Population: Evaluable population included all participants enrolled in the Phase 1b who received at least 1 full dose of MEDI-573, received sorafenib treatment per standard practice during the DLT evaluation period, and completed safety follow-up through the DLT evaluation period or experienced any DLTs during the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

2. Primary Outcome: Phase 1b: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A serious adverse event (SAE) is an AE that results in death, initial or prolonged inpatient hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or an important medical event. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurred first (approximately 15 months).
Time Frame: From the start of study treatment (Day 1) through 60 days after the last dose of MEDI-573 or initiation of another anticancer therapy, whichever occurred first (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
Number analyzed (Participants) | 3 | 3
Participants
  Any TEAEs | 3 | 3
  Any TESAEs | 1 | 1

3. Primary Outcome: Phase 1b: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurred first (approximately 15 months).
Time Frame: as for outcome 2
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
Number analyzed (Participants) | 3 | 3
Participants
  Thrombocytopenia | 2 | 2
  Neutropenia | 1 | 1
  Anemia | 0 | 1
  Blood bilirubin increased | 2 | 2
  Lipase increased | 2 | 1
  Hyperbilirubinemia | 2 | 0
  Aspartate aminotransferase increased | 2 | 0
  Hypophosphataemia | 1 | 1
  Hypoalbuminaemia | 1 | 1
  Alanine aminotransferase increased | 1 | 0
  Amylase increased | 0 | 1
  Blood alkaline phosphatase increased | 1 | 0
  Blood creatinine increased | 0 | 1
  Blood uric acid increased | 0 | 1
  Gamma-glutamyltransferase increased | 1 | 0
  Hypercholesterolaemia | 1 | 0
  Hypocalcaemia | 1 | 0
  Hypoglycaemia | 0 | 1
  Hypomagnesaemia | 1 | 0
  Hematuria | 0 | 1
  Proteinuria | 0 | 1

4. Primary Outcome: Phase 1b: Number of Participants With Vital Signs Abnormalities Reported as TEAEs
Description: An abnormal vital signs that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurred first (approximately 15 months).
Time Frame: as for outcome 2
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
Number analyzed (Participants) | 3 | 3
Participants
  Hypertension | 0 | 2
  Pyrexia | 0 | 1
  Diastolic hypertension | 0 | 1

5. Primary Outcome: Phase 1b: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as TEAEs
Description: An abnormal ECG findings that were judged by the investigator to be medically significant were reported as AEs. The TEAEs are defined as AEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug, up to 60 days after the last study drug or until the participants started another anticancer therapy, whichever occurred first (approximately 15 months).
Time Frame: as for outcome 2
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

6. Primary Outcome: Phase 2: Time to Progression
Description: Phase 2 part of the study was not launched by the sponsor due to strategic business reasons. Therefore, this outcome was not evaluated.
Time Frame: From Day 1 until documentation of progressive disease (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Groups:
- Phase 2 Arm 1: Participants were planned to receive the recommended dose of MEDI-573 from Phase 1b IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
Arm/Group | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI-573
Description: Participants with positive ADA to MEDI-573 are reported in the below table. This outcome was not evaluated for Phase 2 as it was not launched by the sponsor due to strategic business reasons.
Time Frame: Predose on Day 1 of every treatment cycle; end of treatment; Days 30, 60 and 90 post treatment; every 3 months post treatrment till end of study (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 3 | 3 | 0 | 0
Participants | 0 | 0 |  |

8. Secondary Outcome: Phase 2: Best Overall Tumor Response
Description: as for outcome 6
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Arm/Group | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Phase 2: Objective Response Rate
Description: as for outcome 6
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Groups:
- Phase 2 Arm 1: In Phase 2, participants was planned to receive the recommended dose of MEDI-573 from Phase 1b IV on Day 1 of each 21-day cycle and sorafenib 400 mg orally twice daily (Arm 1) or sorafenib 400 mg orally twice daily (Arm 2) until unacceptable toxicity, documentation of disease progression, initiation of alternative anticancer treatment, or withdrawal for other reasons.
Arm/Group | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: as for outcome 6
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Arm/Group | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Phase 2: Change in Tumor Size
Description: Phase 2 part the study was not launched by the sponsor due to strategic business reasons. Therefore, this outcome was not evaluated.
Time Frame: From Day 1 until disease progression or death due to any cause, whichever occurred first (approximately 15 months)
Population: Safety population included all participants who received any amount of study treatment.
Arm/Group | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Phase 1b and Phase 2: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI-573 for Cycle 1
Description: The tmax is defined as actual sampling time to reach maximum observed serum concentration of the study drug. This outcome was not evaluated for Phase 2 as it was not launched by the sponsor due to strategic business reasons.
Time Frame: Cycle 1 (pre-dose; and 5 minutes, 24 hours, Day 8, and Day 15 post-dose); and Cycle 2 Day 1 (pre-dose)
Population: Safety population included all participants who received any amount of study treatment.
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 3 | 3 | 0 | 0
Hours | 1.05 [1.05 to 1.08] | 1.55 [1.52 to 1.58] |  |

13. Secondary Outcome: Phase 1b and Phase 2: Maximum Observed Serum Concentration (Cmax) of MEDI-573 for Cycle 1
Description: The Cmax is the maximum observed serum concentration of study drug. This outcome was not evaluated for Phase 2 as it was not launched by the sponsor due to strategic business reasons.
Time Frame: Cycle 1 (pre-dose; and 5 minutes, 24 hours, Day 8, and Day 15 post-dose); and Cycle 2 Day 1 (pre-dose)
Population: Safety population included all participants who received any amount of study treatment.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 3 | 3 | 0 | 0
mcg/mL | 195 (11.4) | 920 (145) |  |

14. Secondary Outcome: Phase 1b and Phase 2: Area Under Serum Concentration-time Curve From Time Zero to Day 22 (AUC0-Day22) of MEDI-573 for Cycle 1
Description: Area under the concentration-time curve from time zero to Day 22 is reported. This outcome was not evaluated for Phase 2 as it was not launched by the sponsor due to strategic business reasons.
Time Frame: Cycle 1 (pre-dose; and 5 minutes, 24 hours, Day 8, and Day 15 post-dose); and Cycle 2 Day 1 (pre-dose)
Population: Safety population included all participants who received any amount of study treatment.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B | Phase 2 Arm 1 | Phase 2 Arm 2
Number analyzed (Participants) | 3 | 3 | 0 | 0
day*mcg/mL | 887 (231) | 6390 (1440) |  |

ADVERSE EVENTS:
Time Frame: All AEs were reported during safety follow-up period (from the start of study treatment [Day 1] through 60 days after the last dose of MEDI-573 or initiation of another anticancer therapy, whichever occurred first) (approximately 15 months).
Arm/Group | Phase 1b Cohort A | Phase 1b Cohort B
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort A (N=3) | Phase 1b Cohort B (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort A (N=3) | Phase 1b Cohort B (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (10) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Scleral haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 2 (2)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (4)
Implant site pain (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (5) | 0 (0)
Lipase increased (Investigations) | 2 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Diastolic hypertension (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Phase 2 part of the study was not launched by the sponsor due to strategic business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.